CLINICAL TRIAL: NCT05130944
Title: Integrating Psychosocial Support Into Protection and Community Programs for Women in Ecuador and Panama
Brief Title: Feasibility of Community Psychosocial Intervention for Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Copenhagen (Other); HIAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT7637; AID-OAAA17-00002 (Other Grant/Funding Number: United States Agency for International Development)
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Mental Health Wellness 1; Psychological Distress; Coping Skills; Stress
MeSH Terms: interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: Cluster randomized comparative feasibility trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entre Nosotras (group psychosocial intervention) + stress management intervention (Experimental): Experimental condition: Women residing in the study community (displaced and host population) will receive both group psychosocial intervention and stress management intervention. Participants will be given the Spanish version of the Doing What Matters in Times of Stress illustrated guide, that is published and made publicly available by the World Health Organization.
  Interventions: Behavioral: Entre Nosotras; Behavioral: Doing What Matters in Times of Stress
- Entre Nosostras (group psychosocial intervention) (Active Comparator): Comparison condition: Women residing in the study community (displaced and host population) will receive group psychosocial intervention only.
  Interventions: Behavioral: Entre Nosotras

INTERVENTIONS:
Behavioral: Entre Nosotras — A series of five 2-hour group sessions that are administered weekly by two trained female peer facilitators, who are selected by HIAS outreach workers and/or community leaders. The content of the sessions is based on the principles of Psychological First Aid and the Participatory Action Cycle, which is intended to generate community-led problem solving around priority issues affecting their wellbeing.
  Entre Nosotras is a community- and strengths-based intervention designed to mobilize social support, strengthen community connectedness, and stimulate collective action to promote the safety and wellbeing of women.
Behavioral: Doing What Matters in Times of Stress — The stress management components are derived from the World Health Organization Doing What Matters in Times of Stress illustrated guide for coping with adversity (World Health Organization, 2020). The illustrated guide and accompanying audio files are publicly available: https://www.who.int/publications/i/item/9789240003927. During five sessions, the intervention involves 15-20 minute exercises covering a range of stress management and coping skills.
  Other Names: Stress management, coping skills
  Arms: Entre Nosotras (group psychosocial intervention) + stress management intervention

SUMMARY:
The purpose of the current protocol is to describe a cluster randomized feasibility trial examining the integration of a scalable stress management intervention into Entre Nosotras ('among/between us'), a community-based psychosocial intervention for migrant and host community women in Ecuador and Panamá.

Specifically the study aims to:

1. Explore the relevance, acceptability, and feasibility of integrating a stress management intervention into community-based participatory women's group
2. Examine the feasibility of conducting a fully-powered cluster randomized controlled trial evaluating the effectiveness and implementation of integrating a stress management intervention into a community-based participatory women's group as compared to community-based participatory women's groups alone.

DETAILED DESCRIPTION:
The proposed research directly targets two public health areas with major gaps in evidence in the field of humanitarian settings: (1) protection and safety, and (2) mental health and psychosocial wellbeing.

This research will be conducted in three sites in Ecuador and Panama. Latin America has recently experienced increasing levels of forced migration due to political conflict, community violence, and other factors. Panamá and Ecuador host refugees, asylum seekers, and migrants from a range of Central and South American countries (e.g., Colombia, Nicaragua, Venezuela). Migrants in these contexts face mental health and psychosocial problems, threats to their safety, and disrupted social support systems. Gaps in psychosocial services to address these problems despite their high prevalence persist in both countries and have been exacerbated due to the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years) women residing in the study community who speak and understand Spanish
* Displaced or host community members

Exclusion Criteria:

* Severe psychological distress (Kessler-6 >=13)
* Moderate or high risk of suicide
* Cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 275 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Proportion of women screened who are eligible to participate | Baseline
  This is to measure relevance of the intervention in the source population. Appropriateness of the intervention to population needs will be measured using quantitative indicators and qualitative reports from participants and facilitators during the process evaluation.
Proportion of eligible and enrolled women who engage in sessions and/or complete all five group sessions. | Up to 5 weeks
  This is to measure the acceptability of the intervention. Safety, an indicator of acceptability, will also be assessed by adverse events reported during study period. Qualitative interviews with participants and facilitators will inquire about acceptability and will be integrated with quantitative estimates of intervention engagement and completion.
Intervention Usability Scale Score | 5 weeks
  Usability will be measured using the 10-item Intervention Usability Scale, which will be completed by facilitators after the final session of the intervention. Scores are scaled to range from 0-100 with scores exceeding 68 considered to indicate usable interventions.
Recruitment rate | Study period
  The number of individuals enrolled per month will be used to determine the feasibility of a fully-powered definitive trial.
Number of baseline imbalances between study conditions | Baseline
  The number of socio-demographic or study outcome imbalances between the intervention and comparison condition will be used to determine the feasibility of a fully-powered definitive trial and the success of the randomization process.
Attrition - proportion of enrolled individuals who drop out of the study | Up to 10 weeks
  The proportion of enrolled individuals who drop out of the study will be used to indicate the feasibility of a fully-powered definitive trial.
Contamination - proportion of sessions that did not include coping skills intervention components | Up to 5 weeks
  The proportion of experimental sessions that did not include coping skills intervention components and the proportion of control sessions that did include coping skills intervention components from the Doing What Matters in Times of Stress intervention.
Fidelity checklist score | Up to 5 weeks
  Average level of compliance with the intervention activities as intended within the manual. Assessed using a fidelity checklist with average item scores ranging from 0 = not implemented to 2 = implemented well. Scores between 0 and 2 indicate that the activities were partially implemented and/or could be improved.
Facilitator competence score | Up to 5 weeks
  This is to measure the feasibility of the intervention. Facilitator competencies assessed using items from ENACT along qualitative interviews with facilitators will be assessed together. For the quantitative items, we selected six domains that are each scored on a scale from 1=needs improvement to 3=done well.

SECONDARY OUTCOMES:
Personal Wellbeing Index | Baseline, Post-Intervention (approximately 5 Weeks), 5 Weeks Post-Intervention (approximately 10 Weeks)
  This is to measure psychosocial wellbeing; Subscales include satisfaction with standard of living, health, life achievement, personal relationships, personal safety, community connectedness, and future security.
  Each of the nine items is measured on a 0-to-10 scale (0 = No satisfaction at all; 10 = Very satisfied).
Kessler 6 scale score | Baseline, Post-Intervention (approximately 5 Weeks), 5 Weeks Post-Intervention (approximately 10 Weeks)
  This is to measure psychological distress. The Kessler 6 includes six items measured on 5-point Likert scale where respondents indicate the frequency they have experienced a given symptom (from none of the time to all of the time).
Brief COPE scale score | Baseline, Post-Intervention (approximately 5 Weeks), 5 Weeks Post-Intervention (approximately 10 Weeks)
  This is to measure coping. The 28-item scale rates the frequency of using certain coping skills on a 4-point Likert scale from "I haven't been using this at all" to "I've been doing this a lot".
WHODAS Score | Baseline, Post-Intervention (approximately 5 Weeks), 5 Weeks Post-Intervention (approximately 10 Weeks)
  This is to measure functioning. This 12-item scale rates the difficulty individuals have had completing certain tasks on a 5-point Likert Scale from "none" to "extreme or cannot do"
Oslo Social Support Scale Score | Baseline, Post-Intervention (approximately 5 Weeks), 5 Weeks Post-Intervention (approximately 10 Weeks)
  This is to measure social support. This 3-item measure assesses different domains of social support on a 5-point Likert scale with higher values indicating greater levels of social support. Response options vary by item.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Greene, PhD, Principal Investigator — Columbia University
Locations (2):
- HIAS, Quito, Ecuador
- HIAS, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greene MC, Bonz A, Cristobal M, Vega C, Andersen LS, Angulo A, Armijos A, Guevara ME, Benavides L, de la Cruz A, Lopez MJ, Moyano A, Murcia A, Noboa MJ, Rodriguez A, Solis J, Vergara D, Scharf J, Dutt P, Wainberg M, Tol WA. Evaluating the feasibility of a group psychosocial intervention for migrant and host community women in Ecuador and Panama: protocol for a multi-site feasibility cluster trial. Pilot Feasibility Stud. 2022 Jun 15;8(1):126. doi: 10.1186/s40814-022-01085-1. PMID 35706068